CLINICAL TRIAL: NCT05851833
Title: A Retrospective Study of Early Postoperative Mobilization in the Recovery of Patients With Oral Head and Neck Tumors Who Underwent Flap Reconstruction
Status: Completed | Type: Observational
Sponsor: Jie He, MD (Other)
Responsible Party: Sponsor-Investigator, Jie He, MD, Associate chief physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Other Study IDs: 654321
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Length of Hospital Stay
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early MobilizatioN
  Interventions: Behavioral: Early Mobilization
- conventional Mobilization

INTERVENTIONS:
Behavioral: Early Mobilization — The time the patient began to sit, stand, and walk after surgery is earlier than traditional model.
  Groups: Early MobilizatioN

SUMMARY:
All patients with head and neck cancers and osteomyelitis who underwent vascularized flap reconstruction at Shanghai Ninth People's Hospital (North Campus), Shanghai Jiao Tong University, from February 2020 to July 2021 were the object of a retrospective data collection.Depending on whether they had postoperative early mobilization, all patients were split into experimental and control groups.In the experimental group, patients were split into two groups based on the postoperative day(POD): the POD 0-1 group and the POD >1 group.Comparison and analysis were done on the difference in hospital days and post-operative complication rates between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with head and neck diseases undergoing flap reconstruction and repair
2. Patients with complete data preservation and consent
3. Patients who follow medical advice during hospitalization

Exclusion Criteria:

1. Patients who survived less than 1 month after surgery
2. Patients with other tumors before surgery 3, mental patients, audio-visual impairment or uncooperative patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Early Mobilizationon Recovery After Major Head and Neck Surgery With Flap Reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay after surgery | February 2020 to July 2021
  The time span between the end of surgery and hospital discharge is defined as the length of hospital stay after surgery.

SECONDARY OUTCOMES:
pulmonary infection rate | February 2020 to July 2021
  The pulmonary infection rate is calculated as the proportion of hospitalized patients who had pulmonary infections over all patients.
deep vein thrombosis rate | February 2020 to July 2021
  The deep vein thrombosis rate is calculated as the proportion of hospitalized patients who had deep vein thrombosis over all patients.
flap crisis rate | February 2020 to July 2021
  The flap crisis rate is calculated as the proportion of hospitalized patients who had flap crisis over all patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China